CLINICAL TRIAL: NCT05726513
Title: Evaluation of Regional Ventilation Distribution Using Electrical Impedance Tomography During Weaning From Mechanical Ventilation
Acronym: WEAN-EIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Università degli Studi di Ferrara (Other)
Collaborators: University of Milan (Other)
Responsible Party: Principal Investigator, Savino Spadaro, Principal investigator, Università degli Studi di Ferrara
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: WEAN-EIT
Record Dates: First submitted 2023-01-13; First posted 2023-02-14 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Acute Respiratory Failure; Mechanical Ventilation Complication; Ventilator-Induced Lung Injury; Weaning Failure
Keywords: Electrical Impedance tomography; Weaning trial; Acute respiratory failure; Lung monitoring
MeSH Terms: conditions — Ventilator-Induced Lung Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low support, high Positive end-expiratory pressure (Other): Low support, high Positive end-expiratory pressure
  Interventions: Diagnostic Test: Weaning trial - Low support, high Positive end-expiratory pressure
- Low support, zero positive end-expiratory pressure (Other): Low support, zero positive end-expiratory pressure
  Interventions: Diagnostic Test: Weaning trial - Low support, zero positive end-expiratory pressure
- Zero support, zero positive end-expiratory pressure (Other): Zero support, zero positive end-expiratory pressure
  Interventions: Diagnostic Test: Weaning trial - Zero support, zero positive end-expiratory pressure

INTERVENTIONS:
Diagnostic Test: Weaning trial - Low support, high Positive end-expiratory pressure — The researcher will evaluate the readiness to be weaned of the patient using a weaning trial with low pressure support ventilation and a positive end expiratory pressure of 5 cmH2O
  Arms: Low support, high Positive end-expiratory pressure
Diagnostic Test: Weaning trial - Low support, zero positive end-expiratory pressure — The researcher will evaluate the readiness to be weaned of the patient using a weaning trial with low pressure support ventilation and a positive end expiratory pressure of 0 cmH2O
  Arms: Low support, zero positive end-expiratory pressure
Diagnostic Test: Weaning trial - Zero support, zero positive end-expiratory pressure — The researcher will evaluate the readiness to be weaned of the patient using a weaning trial with 0 pressure support ventilation and a positive end expiratory pressure of 0 cmH2O
  Arms: Zero support, zero positive end-expiratory pressure

SUMMARY:
The goal of this physiological cross-over clinical trial is to evaluate the effect of different clinically used weaning trials on regional mechanical ventilation in a population of patients undergoing weaning from mechanical ventilation for acute respiratory failure.

The main question[s] it aims to answer are:

* to evaluate which weaning trial is associated to a better regional ventilation distribution
* to evaluate which weaning trial can be comparable to ventilation distribution after extubation

Participants will undergo 3 clinically used weaning trials in a random order (cross-over trial). Researchers will compare the different steps to see if regional ventilation distribution is different among the different trial .

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 and < 70 years
* Ready to be weaned from mechanical ventilation according to clinical criteria

Exclusion Criteria:

* Age < 18 years or > 70 years
* Presence of chest drains
* Presence of pacemaker/impantable cardiac device;
* diagnosis of Pneumothorax, or pneumomediastinum
* Diagnois of neuromuscular diseases
* Use of neuromuscular blockers in the 48 hours before screening;
* Body mass index > 35 kg/m2
* Refusal to participate of the patient/next of kin

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-02-15 (Estimated); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Regional Ventilation distribution using Electrical Impedance Tomography | 2 hours
  The researchers will evaluate differences in ventilation distribution pattern among the different weaning trials using Electrical Impedance Tomography and focusing on:
  * Regional ventilation distribution
  * Regional inhomogeneity
  * Regional compliance distribution
  * Center of Ventilation
  * Silent Spaces

SECONDARY OUTCOMES:
Differences in Regional Ventilation distribution using Electrical Impedance Tomography between weaning trials and post-extubation phase | 48 hours
  The researchers will evaluate differences in ventilation distribution pattern among the different weaning trials and the post-extubation phase using Electrical Impedance Tomography and focusing on:
  * Regional ventilation distribution
  * Regional inhomogeneity
  * Regional compliance distribution
  * Center of Ventilation
  * Silent Spaces

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliero Universitaria Sant'Anna, Ferrara, Italy

IPD SHARING:
Plan to Share IPD: No